CLINICAL TRIAL: NCT03272776
Title: A Multicenter Study of the Protector Laryngeal Mask in Non Paralyzed, Anesthetized Patients
Brief Title: Multicenter Study of the Protector Laryngeal Mask
Status: Completed | Type: Observational
Sponsor: Matilde Zaballos (Other)
Collaborators: Teleflex (Industry)
Responsible Party: Sponsor-Investigator, Matilde Zaballos, Anesthesiologist, Hospital General Universitario Gregorio Marañon
Organization: Hospital General Universitario Gregorio Marañon (Other)
Other Study IDs: MASKAPROTECTOR
Record Dates: First submitted 2017-08-22; First posted 2017-09-06 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Airway
Keywords: LMA Protector; Second Generation Laryngeal Masks; Airway; Dual Gastric Acces; Teleflex; Supraglottic Devices; Ambulatory Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Protector Laryngeal Mask Airway: Patients undergoing anesthesia in which airway management includes a Protector Laryngeal Mask and fulfill the inclusion criteria of the study.
  Interventions: Device: Protector Laryngeal Mask airway

INTERVENTIONS:
Device: Protector Laryngeal Mask airway — Evaluate the time of insertion, performance, security and insertion success rate of the Protector Laryngeal Mask in patients under general anasthesia.

SUMMARY:
The study was designed to evaluate the success rate, time of insertion, sealing efficacy and security of the Protector Laryngeal Mask, a new second generation disposable supraglottic airway device, in patients undergoing elective surgery.

DETAILED DESCRIPTION:
Laryngeal masks (LM) and supraglottic devices (SGD), in all their different forms, have become an authentic innovation in airway management especially in day surgery.

LMA Protector (Teleflex Medical, Athlone, Ireland) is a new disposable SGD currently available for anaesthetic practice. It is made of silicone (with no latex in its composition) and shares some of the characteristics of the second generation SGDs (as the presence of a gastric access channel); however, it has an additional drainage channel, both channels terminate distally in a camera behind the mask cuff. The presence of two drainage channels ("male" and "female") increases the patient safety against regurgitation, both of distal gastric content and secretions located in the oropharyngeal region. The gastric access channel called "female" also allows the insertion of a nasogastric tube if required. These drainage channels are useful for diagnosing the correct position of the mask, since the observation of leaks or gas through it can help diagnose a displacement the mask.

LMA Protector is designed with a preformed anatomic curve, and the airway conduct has an elliptical cross section, which ends distally in the mask. This design follows the anatomy of the human airway, which facilitates the insertion of the device. The softness of the mask material allows easy insertion.

Doubts regarding the transmission of infectious diseases with reusable devices makes disposable devices such as LMA Protector, one of the most interesting devices for use in anaesthetic procedures that are usually performed with SGD.

Its characteristics in the design, composition by a smooth and atraumatic material, the presence of two gastric drainage accesses, with potential improved patient safety and its characteristic of being disposable suggests a significant expansion of its use in the coming years .

In contrast to other SGDs that have been evaluated extensively, to date there are no large clinical studies showing its suitably and performance in a daily clinical scenario.

ELIGIBILITY:
Inclusion Criteria:

* Surgery procedures usually performed with supraglottic devices.
* ASA physical status I-III patients
* Age 18-75
* Signed inform consent

Exclusion Criteria:

* Patients with known difficult airway
* Patients with predicted difficult airway
* Patients with increased risk of aspiration
* Patient refusal to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing surgery procedures in any of the collaborating centers of the study that fulfill the inclusion and exclusion criteria described below.
Sampling Method: Non-Probability Sample
Enrollment: 280 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Evaluate the number of attempts to insert of the LMA Protector | The number of insertion attempts will be collected after anesthesia induction: 1 minute after the administration of propofol
  Insertion attempts: from picking up the LMA Protector until the mask is placed into the patient mouth . (in numbers)

SECONDARY OUTCOMES:
Blood pressure during insertion of LMA protect | Baseline and every 3 minutes until 6 minutes after insertion of the LMA protector
  Blood pressure in mmHg
Heart rate during insertion of LMA protect | Baseline and every 3 minutes until 6 minutes after insertion of the LMA protector
  heart rate in beep per minute
BIS data | Baseline and every 3 minutes until 6 minutes after insertion of the LMA protector (To evaluate the evolution of BIS values during insertion of the LMA
  number from 100 (awake) to 40-45 (anesthetic status)
Oropharyngeal leak pressure of the LMA Protector | The Oropharyngeal leak pressure of the LMA Protector will be collected 5 minutes after the LMA Protector will be inserted
  The Oropharyngeal leak pressure of the LMA Protector will be determined with an intracuff pressure of 60 cm H2O by closing the expiratory valve of the breathing circle circuit at a fixed gas flow of 3 L/min and noting the pressure at which an oropharyngeal leak occurs. (in cm H2O)

CONTACTS AND LOCATIONS:
Overall Officials: Maite López-Gil, Study Chair — Servicio de Anestesiología, Hospital General Universitario Gregorio Marañon
Locations (1):
- Servicio de Anestesia, Hospital General Universitario Gregorio Marañon, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brimacombe JR, editor. Laryngeal Mask Anesthesia. Principles and practice. 2nd Ed. Filadelfia. 2005.
- [Background] Van Zundert AA, Skinner MW, Van Zundert TC, Luney SR, Pandit JJ. Value of knowing physical characteristics of the airway device before using it. Br J Anaesth. 2016 Jul;117(1):12-6. doi: 10.1093/bja/aew106. Epub 2016 May 4. No abstract available. PMID 27147543
- [Background] Zaballos García M, López Álvarez S, Agustí Martínez-Marcos S, Blanco Sánchez T, Bustos Molina F, Cabré Fabré P, et al. Nuevas aportaciones de la mascarilla laríngea en cirugía ambulatoria. Contribución de la mascarilla laríngea Supreme. Cir May Amb 2011; 16(2): 60-6.
- [Background] Zaballos García M, López Álvarez S, Agustí Martínez-Marcos S, Blanco Sánchez T, Bustos Molina F, Cabré Fabré P, Cordero Lorenzo JM, Izquierdo Villaroya B, Lafuente Ojeda N, M. López Gil M, Rodríguez Archilla A, Zaballos Bustingorri J Recomendaciones prácticas de uso de la mascarilla laríngea en Cirugía Ambulatoria. Cir May Amb 2008; 13: (1) 4-26.